CLINICAL TRIAL: NCT01210196
Title: Sophisticated Assessment of Disease Burden in Patients With Fabry Disease - The SOPHIA in Fabry Disease Study
Brief Title: Sophisticated Assessment of Disease Burden in Patients With Fabry Disease
Acronym: SOPHIA
Status: Completed | Type: Observational
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: Shire/CS01
Record Dates: First submitted 2010-09-25; First posted 2010-09-28 (Estimated); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Fabry Disease
Keywords: Fabry
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- mild affected Fabry patients
  Interventions: Procedure: MRI

INTERVENTIONS:
Procedure: MRI — Cardiac MRI after 12 and 24 months.
  Other Names: MRT (German)

SUMMARY:
To detect early signs of cardiac and metabolic alterations as well as to evaluate the progression of cardiac and metabolic impairments in mildly affected patients with Fabry Disease using high sensitive diagnostic methods.

DETAILED DESCRIPTION:
Observational Study Evaluating the use of cardiac MRI with late enhancement technique, Echocardiography, 24h Holter ECG, plasma Lyso-Gb3 and urinary Gb3, to identify early signs of progressive Fabry Disease.

ELIGIBILITY:
Inclusion Criteria:

1. Women: A confirmed exonic mutation within the α-Galactosidase gene Men: A confirmed exonic mutation within the α-Galactosidas gene and/or reduced α- Galactosidase activity
2. Female patients ≥ 25 years-old and male patients ≥ 25 years-old
3. The patient has not received enzyme replacement therapy for treatment of Fabry disease
4. The patient must have voluntarily signed an Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved informed consent form after all relevant aspects of the study have been explained and discussed with the patient
5. The patient has already mild symptoms of Fabry disease presented in at least one minor organ involvement, e.g. proteinuria 1, mild cardiac symptoms not needing treatment yet, pain attacks, gastrointestinal symptoms or history of TIA.

Exclusion Criteria:

1. The patient has received ERT or investigational product(s) for any reason within 30 days prior to study entry.
2. Any contraindication for MRI-diagnosis
3. Incompatibility to MRI contrast agent (elevated serum creatinine - according to SPC of contrast medium) The patient is unable to comply with the protocol, e.g., has a clinically relevant medical condition making implementation of the protocol difficult; has an uncooperative attitude; is unable to return for study evaluations; or is otherwise unlikely to complete the study, as determined by the investigator.
4. Planned ERT within the next 24 months (nevertheless if a ERT becomes medically necessary in the observational period ERT might be introduced)

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients with a genetically confirmed Fabry disease.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2010-10-31 (Actual); Primary Completion 2013-09-30 (Actual); Study Completion 2013-09-30 (Actual)

PRIMARY OUTCOMES:
Number of fibrotic left ventricular segments at baseline and after 12 and 24 months | 24 months

SECONDARY OUTCOMES:
Left ventricular mass at 12 and 24 months compared to baseline assessed by MRI | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (11):
- Belgium (2):
  - ZNA Middelheim, Antwerp
  - Institute of Pathology et de Génétique (IPG), Gosselies
- Charles University in Prague and General University Hospital in Prague, Prague, Czechia
- National University Hospital, Rigshospitalet, Copenhagen, Denmark
- Turku University Hospital, Turku, Finland
- Germany (5):
  - Charité University Medicine Campus Mitte, Berlin
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - University of Mainz, Mainz
  - University Hospital of Münster, Münster
  - University Hospital Würzburg, Würzburg
- Uppsala University Hospital, Uppsala, Sweden

REFERENCES:
- [Derived] Weidemann F, Beer M, Kralewski M, Siwy J, Kampmann C. Early detection of organ involvement in Fabry disease by biomarker assessment in conjunction with LGE cardiac MRI: results from the SOPHIA study. Mol Genet Metab. 2019 Feb;126(2):169-182. doi: 10.1016/j.ymgme.2018.11.005. Epub 2018 Nov 12. PMID 30594474